CLINICAL TRIAL: NCT05501665
Title: SiCARIO (Split Course Adaptive Radioimmunotherapy) for the Treatment of Oligometastatic Non-Small Cell Lung Cancer (NSCLC) Using Biologically-Adaptive Radiotherapy - A Phase I/II Study
Brief Title: Split Course Adaptive Radiation Therapy With Pembrolizumab With/Without Chemotherapy for Treating Stage IV Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Evan Osmundson, MD, PhD, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICCTHOP2185; NCI-2022-05101 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICCTHOP2185 (Other: Vanderbilt University/Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage III Lung Cancer
Keywords: Oligometastasis; Adaptive Radiotherapy; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; Carboplatin; Fluorodeoxyglucose F18; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; pembrolizumab; Pemetrexed; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Fluorine-18; 4-(3-fluoropropyl)glutamic acid; Ipilimumab; Nivolumab; cemiplimab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (11):
- Arm 1 (carboplatin, pemetrexed, pembrolizumab, radiation) (Experimental): Patients receive carboplatin, pemetrexed, and pembrolizumab on day 1 of each cycle. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pemetrexed and pembrolizumab on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Biological: Pembrolizumab; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan
- Arm II (carboplatin, pemetrexed, cemiplimab, radiation) (Experimental): Patients receive carboplatin, pemetrexed and cemiplimab-rwlc on day 1 of each cycle. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pemetrexed and cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan; Biological: Cemiplimab
- Arm III (carboplatin, paclitaxel, cemiplimab-rwlc, radiation) (Experimental): Patients receive carboplatin, paclitaxel and cemiplimab-rwlc on day 1 of each cycle. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pemetrexed and cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Nab-paclitaxel; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan; Biological: Cemiplimab
- Arm IV (Carbo, pemetrexed, nivolumab, ipilimumab, radiation) (Experimental): Patients receive carboplatin, pemetrexed and nivolumab on day 1 of each cycle and ipilimumab on day 1 of every other cycle. Treatment repeats for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then continue to receive ipilmumab and nivolumab on the same schedule for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan; Biological: Ipilimumab; Biological: Nivolumab
- Arm V (Carboplatin, paclitaxel, pembrolizumab, radiation) (Experimental): Patients receive carboplatin, paclitaxel, and pembrolizumab on day 1 of each cycle. Treatment repeats every 3 weeks for 4 up to cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. Patients then receive pembrolizumab on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Nab-paclitaxel; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan
- Arm VI (Carboplatin, paclitaxel, cemiplimab-rwlc, radiation) (Experimental): Patients receive carboplatin, paclitaxel, and cemiplimab-rwlc on day 1 of each cycle. Treatment repeats every 3 weeks for 4 up to cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. Patients then receive cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Nab-paclitaxel; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan; Biological: Cemiplimab
- Arm VII (carbo, paclitaxel, nivolumab, ipilimumab, radiation) (Experimental): Patients receive carboplatin, paclitaxel, and cemiplimab-rwlc on day 1 of each cycle. Treatment repeats every 3 weeks for 4 up to cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. Patients then receive cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Nab-paclitaxel; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan; Biological: Ipilimumab; Biological: Nivolumab
- Arm VIII (pembrolizumab, radiation) (Experimental): Patients receive pembrolizumab on day 1 of each cycle. Cycles repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan
- Arm IX (atezolizumab, radiation) (Experimental): Patients receive atezolizumab on day 1 of each cycle. Cycles repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan; Biological: Atezolizumab
- Arm X (cemiplimab-rwlc, radiation) (Experimental): Patients receive cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.
  All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan; Biological: Cemiplimab
- Arm XI (nivolumab, ipilumumab, radiation) (Experimental): Patients receive ipilmumab every 6 weeks and nivolumab every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan; Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given carboplatin
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm 1 (carboplatin, pemetrexed, pembrolizumab, radiation); Arm II (carboplatin, pemetrexed, cemiplimab, radiation); Arm III (carboplatin, paclitaxel, cemiplimab-rwlc, radiation); Arm IV (Carbo, pemetrexed, nivolumab, ipilimumab, radiation); Arm V (Carboplatin, paclitaxel, pembrolizumab, radiation); Arm VI (Carboplatin, paclitaxel, cemiplimab-rwlc, radiation); Arm VII (carbo, paclitaxel, nivolumab, ipilimumab, radiation)
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Nab-paclitaxel — Given nab-paclitaxel
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
  Arms: Arm III (carboplatin, paclitaxel, cemiplimab-rwlc, radiation); Arm V (Carboplatin, paclitaxel, pembrolizumab, radiation); Arm VI (Carboplatin, paclitaxel, cemiplimab-rwlc, radiation); Arm VII (carbo, paclitaxel, nivolumab, ipilimumab, radiation)
Biological: Pembrolizumab — Given pembrolizumab
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm 1 (carboplatin, pemetrexed, pembrolizumab, radiation); Arm V (Carboplatin, paclitaxel, pembrolizumab, radiation); Arm VIII (pembrolizumab, radiation)
Drug: Pemetrexed — Given pemetrexed
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
  Arms: Arm 1 (carboplatin, pemetrexed, pembrolizumab, radiation); Arm II (carboplatin, pemetrexed, cemiplimab, radiation); Arm IV (Carbo, pemetrexed, nivolumab, ipilimumab, radiation)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Other: [18-F] (fluoropropyl)-L-glutamate (FSPG) PET scan — Undergo PET scan
Biological: Ipilimumab — Given Ipilimumab
  Arms: Arm IV (Carbo, pemetrexed, nivolumab, ipilimumab, radiation); Arm VII (carbo, paclitaxel, nivolumab, ipilimumab, radiation); Arm XI (nivolumab, ipilumumab, radiation)
Biological: Nivolumab — Given Nivolumab
  Arms: Arm IV (Carbo, pemetrexed, nivolumab, ipilimumab, radiation); Arm VII (carbo, paclitaxel, nivolumab, ipilimumab, radiation); Arm XI (nivolumab, ipilumumab, radiation)
Biological: Cemiplimab — Given Cemiplimab
  Arms: Arm II (carboplatin, pemetrexed, cemiplimab, radiation); Arm III (carboplatin, paclitaxel, cemiplimab-rwlc, radiation); Arm VI (Carboplatin, paclitaxel, cemiplimab-rwlc, radiation); Arm X (cemiplimab-rwlc, radiation)
Biological: Atezolizumab — Given Atezolizumab
  Arms: Arm IX (atezolizumab, radiation)

SUMMARY:
This phase I/II trial tests the safety and efficacy of split-course adaptive radiation therapy in combination with immunotherapy with or without chemotherapy for the treatment of patients with stage IV lung cancer or lung cancer that that has spread to nearby tissue or lymph nodes (locally advanced). Radiation therapy is a standard cancer treatment that uses high energy rays to kill cancer cells and shrink tumors. Split-course adaptive radiation therapy uses patient disease response to alter the intensity of the radiation therapy. Immunotherapy with monoclonal antibodies such as pembrolizumab, ipilimumab, cemiplimab, atezolizumab or nivolumab may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs like carboplatin, pemetrexed, and paclitaxel work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving split-course adaptive radiation therapy with standard treatments like immunotherapy and chemotherapy may be more effective at treating stage IV or locally advanced lung cancer than giving them alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of adaptive split course hypo-fractionated radiation therapy (RT) with immunotherapy containing systemic regimens.

II. Evaluate efficacy of the use of adaptive split course hypo-fractionated RT with immunotherapy containing systemic regimens.

SECONDARY OBJECTIVES:

I. Evaluate progression and survival benefit of split course adaptive radioimmunotherapy (SiCARIO) regimen.

II. Identify potential functional radiomic biomarkers of response to SiCARIO regimen.

III. Develop real-world clinical and treatment planning workflows for implementation of the Ethos platform for anatomic and biologically adaptive RT.

OUTLINE:

PRIMARY OBJECTIVES:

I. Evaluate the safety of adaptive split course hypo-fractionated radiation therapy (RT) with immunotherapy containing systemic regimens.

II. Evaluate efficacy of the use of adaptive split course hypo-fractionated RT with immunotherapy containing systemic regimens.

SECONDARY OBJECTIVES:

I. Evaluate progression and survival benefit of split course adaptive radioimmunotherapy (SiCARIO) regimen.

II. Identify potential functional radiomic biomarkers of response to SiCARIO regimen.

III. Develop real-world clinical and treatment planning workflows for implementation of the Ethos platform for anatomic and biologically adaptive RT.

OUTLINE:

Patients are assigned to 1 of 11 standard treatment regimens, in combination with radiation therapy, as determined by the tumor histology and PD-L1 status.

Patients with non-squamous histology and any PD-L1 status are assigned to arms 1-4.

ARM I: Patients receive carboplatin, pemetrexed, and pembrolizumab on day 1 of each cycle. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pemetrexed and pembrolizumab on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

ARM II: Patients receive carboplatin, pemetrexed and cemiplimab-rwlc on day 1 of each cycle. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pemetrexed and cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

ARM III: Patients receive carboplatin, paclitaxel and cemiplimab-rwlc on day 1 of each cycle. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pemetrexed and cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

ARM IV: Patients receive carboplatin, pemetrexed and nivolumab on day 1 of each cycle and ipilimumab on day 1 of every other cycle. Treatment repeats for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then continue to receive ipilmumab and nivolumab on the same schedule for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

Patients with squamous histology and any PD-L1 histology are assigned to arms 5-7

ARM V: Patients receive carboplatin, paclitaxel, and pembrolizumab on day 1 of each cycle. Treatment repeats every 3 weeks for 4 up to cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. Patients then receive pembrolizumab on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.

ARM VI: Patients receive carboplatin, paclitaxel, and cemiplimab-rwlc on day 1 of each cycle. Treatment repeats every 3 weeks for 4 up to cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions. Patients then receive cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.

ARM VII: Patients receive carboplatin, paclitaxel and nivolumab on day 1 of each cycle and ipilimumab on day 1 of every other cycle. Treatment repeats for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then continue to receive ipilmumab and nivolumab on the same schedule for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

Patients with PD-L1 ≥ 50% are assigned to arms 8-10

ARM VIII: Patients receive pembrolizumab on day 1 of each cycle. Cycles repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

ARM IX: Patients receive atezolizumab on day 1 of each cycle. Cycles repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

ARM X: Patients receive cemiplimab-rwlc on day 1 of each cycle. Cycles repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

Patients with any PD-L1 status or histology who are not a chemotherapy candidate are assigned to arm 11

ARM XI: Patients receive ipilmumab every 6 weeks and nivolumab every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on day 1 of each cycle over 5 treatment fractions.

All patients also receive fludeoxyglucose F-18 intravenously and fluorine F 18 florilglutamic acid IV and undergo PET/ CT during screening and on study. Patients also undergo collection of blood samples, as well as CT and MRI throughout the trial.

After completion of study treatment, patients are followed up at 4 weeks, 12 weeks, and then every 12 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at time of informed consent
* • Histologically documented or cytologically confirmed diagnosis of stage IVA or IVB (M1b or M1c) or locally advanced (not eligible for standard of care [SOC] chemoradiation) non-small cell lung cancer with evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria
* Available tumor material (< 6 months old) adequate for confirmation of programmed cell death 1 ligand 1 (PD-L1) expression per local standard of care testing
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate organ function to receive therapy as determined by investigators and other treating physicians
* Participants with brain metastases that can be comprehensively managed with surgery and/or stereotactic radiosurgery, prior to initiation of chemo-immunotherapy are allowed. Number of brain metastases allowed is not specified at eligibility is at discretion of investigator
* Contraceptive use should be initiated or continued per guidance in labeling for approved chemotherapies
* Female patients must be non-pregnant and not breastfeeding.

  * If woman of childbearing potential (WOCBP), must utilize highly effective contraceptive method (failure rate of < 1% per year) throughout intervention period and continued per guidance specified in labeling for approved chemotherapies. Must have negative pregnancy test (serum or urine) within 1 week prior to initiation of first cycle of therapy
* Eligible for immunotherapy-based systemic regimens per judgment of patient's study physician
* Able to submit written informed consent

Exclusion Criteria:

* Mixed small cell histology
* Confirmed candidate (per study physician) for alternative systemic therapy if preferred by treating physician (i.e. mEGFR, ALK, KRAS G12C or ROS1 mutations). Testing not required for enrollment
* Brain metastases that would require administration of whole brain radiotherapy for management on required screening brain MRI within 21 days of day 1 of study treatment
* Symptomatic malignant ascites or malignant pleural effusion (sampling not required). Pleural metastases are allowed if deemed targetable with radiotherapy
* Major surgery (requiring general anesthesia or at discretion of study physician) within 4 weeks prior to study enrollment that would prevent treatment with SiCARIO regimen
* History of organ transplant requiring therapeutic immunosuppression
* Known clinically significant (per study physician) acute or chronic infections including human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or active tuberculosis (testing not required). Patients with HBV and HCV must be on stable dose of antiviral therapy on study entry
* Uncontrolled intercurrent illness including, but not limited to, New York Heart Association (NYHA) class III-IV congestive heart failure, uncontrolled hypertension (average systolic blood pressure greater than or equal to 140 or average diastolic blood pressure greater than or equal to 90 despite optimal medical therapy), unstable angina pectoris, cardiac arrythmia, active peptic ulcer disease, bleeding diatheses or psychiatric illness that would limit in the judgment of the study physician
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization within 30 days of day 1 of study treatment
* History of prior independent malignancy within 3 years of enrollment, except for adequately treated basal or squamous cell carcinoma of the skin, adequately treated carcinoma in situ (e.g. cervix or non-invasive bladder cancer)
* Receipt of prior >1 cycle of immune checkpoint inhibitor for current malignancy (prior cytotoxic chemotherapy is allowed)
* Prior radiotherapy that would preclude delivery of protocol- based radiotherapy to normal organ tolerance per patient's study physician
* Current or prior use of immunosuppressive medications within 28 days of enrollment with exception of intranasal or inhaled corticosteroids or systemic steroids at physiologic doses (equivalent to less than or equal to 10 mg/day of prednisone). Systemic steroids required during therapy for adverse event (AE) management and for residual neurologic complications from management of central nervous system (CNS) metastases are allowed at doses exceeding 10 mg/day of prednisone equivalents
* Active autoimmune disease requiring systemic treatment within past 1 year
* Receipt of live attenuated vaccine within 30 days of enrollment
* Use of prohibited concomitant drug within 30 days of enrollment
* Known severe (>= grade 3 Common Terminology Criteria for Adverse Events [CTCAE]) hypersensitivity to study intervention or formulation
* Concurrent enrollment in another clinical trial (unless observational or within follow-up period)
* Any condition at discretion of investigator that will preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Safety endpoints will be tabulated using descriptive statistics, and by appropriate subgroups. The incidence of adverse events will be summarized according to organ system in terms of severity by Common Terminology Criteria for Adverse Events and relationship to treatment
Best overall response rate | Within 6 months
  By Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Exact binomial test and 95% confidence interval (CI) will be used.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Time from consent to the date of first documentation of objective progressive disease assessed by RECIST 1.1 or death, assessed at 6, 9, and 12 months
  Estimation of the treatment effect by a Cox proportional hazards model (stratified by chemotherapy regimen and PD-L1 expression, each stratum defines separate baseline hazard function); ties handled by replacing the proportional hazards model by the discrete logistic model; 95% CI for the hazard ratio will be calculated. Kaplan-Meier estimates and associated statistics (PFS rates at 6, 9, 12; median PFS) and corresponding 95% CI will be presented by treatment group.
Overall survival | Time from consent to the date of death due to any cause, assessed up to 2 years
  Estimation of the treatment effect by a Cox proportional hazards model (stratified by chemotherapy regimen and PD-L1 expression, each stratum defines separate baseline hazard function); ties handled by replacing the proportional hazards model by the discrete logistic model; 95% CI for the hazard ratio will be calculated. Kaplan-Meier estimates and associated statistics and corresponding 95% CI will be presented by treatment group.
New metastasis free survival | Time from consent to the date of the first documentation of a new distant metastasis or death, assessed up to 2 years
  Any new lesions different from the ones present at screening are considered as new metastases.
Quantitative and qualitative markers of planning and treatment resource utilization | Up to 2 years
  Develop real-world clinical and treatment planning workflows for implementation of the Ethos platform for anatomic and biologically adaptive radiation therapy (RT).

CONTACTS AND LOCATIONS:
Overall Officials: Evan Osmundson, MD, PhD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT05501665/ICF_000.pdf